CLINICAL TRIAL: NCT00720109
Title: Intensified Tyrosine Kinase Inhibitor Therapy (Dasatinib NSC# 732517) in Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia (ALL)
Brief Title: Dasatinib and Combination Chemotherapy in Treating Young Patients With Newly Diagnosed Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00312; NCI-2009-00312 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AALL0622; CDR0000600217; 08-829; COG-AALL0622; AALL0622 (Other: Childrens Oncology Group); AALL0622 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2008-07-19; First posted 2008-07-22 (Estimated); Results first posted 2016-10-07 (Estimated); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Acute Lymphoblastic Leukemia; Adult B Acute Lymphoblastic Leukemia With t(9;22)(q34.1;q11.2); BCR-ABL1; Childhood B Acute Lymphoblastic Leukemia With t(9;22)(q34.1;q11.2); BCR-ABL1
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase; Leyk; Cyclophosphamide; Cytarabine; Dasatinib; Daunorubicin; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Etoposide; Filgrastim; Granulocyte Colony-Stimulating Factor; Hydrocortisone; hydrocortisone hemisuccinate; Ifosfamide; Leucovorin; Mercaptopurine; azathiopurine; Methotrexate; merphos; Methylprednisolone; exifone; Medrol Veriderm; pegaspargase; Prednisone; deltacortene; prednylidene; Radiotherapy; Radiation; Vincristine

ARMS (1):
- Treatment (enzyme inhibitor therapy and chemotherapy) (Experimental): See Detailed Description
  Interventions: Drug: Asparaginase; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dasatinib; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Drug: Etoposide; Biological: Filgrastim; Drug: Hydrocortisone Sodium Succinate; Drug: Ifosfamide; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Methylprednisolone; Drug: Pegaspargase; Drug: Prednisone; Radiation: Radiation Therapy; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Asparaginase — Given IT
  Other Names: ASP-1; Asparaginase II; Asparaginase-E.Coli; Colaspase; Elspar; Kidrolase; L-Asnase; L-ASP; L-asparaginase; L-Asparagine amidohydrolase; Laspar; Lcf-ASP; Leucogen; Leunase; MK-965; Paronal; Re-82-TAD-15; Serasa; Spectrila
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given IT or IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Dasatinib Hydrate; Dasatinib Monohydrate; Sprycel
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Drug: Dexamethasone — Given IV or PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Biological: Filgrastim — Given IV or SC
  Other Names: G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
Drug: Hydrocortisone Sodium Succinate — Given IT
  Other Names: (11beta)-21-(3-Carboxy-1-oxopropyl)-11,17-dihydroxypregn-4-ene-3,20-dione, Monosodium Salt; A-Hydrocort; Buccalsone; Corlan; Cortisol sodium succinate; Cortop; Efcortelan; Emergent-EZ; Flebocortid; Hidroc Clora; Hycorace; Hydro-Adreson; Hydrocort; Hydrocortisone 21-Sodium Succinate; Hydrocortisone Na Succinate; Kinogen; Nordicort; Nositrol; Sinsurrene; Sodium hydrocortisone succinate; Solu-Cortef; Solu-Glyc
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Leucovorin Calcium — Given IV or PO
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; citrovorum factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; BW 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Methotrexate — Given IT, PO, or IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Methylprednisolone — Given IV
  Other Names: Adlone; Caberdelta M; DepMedalone; Depo Moderin; Depo-Nisolone; Duralone; Emmetipi; Esametone; Firmacort; Medlone 21; Medrate; Medrol; Medrol Veriderm; Medrone; Mega-Star; Meprolone; Methylprednisolonum; Metilbetasone Solubile; Metrocort; Metypresol; Metysolon; Predni-M-Tablinen; Prednilen; Radilem; Sieropresol; Solpredone; Summicort; Urbason; Veriderm Medrol; Wyacort
Drug: Pegaspargase — Given IM
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; Oncaspar-IV; PEG-asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
Drug: Prednisone — Given PO or IV
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Radiation: Radiation Therapy — Some patients undergo cranial RT
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase II/III trial is studying the side effects and how well giving dasatinib together with combination chemotherapy works in treating young patients with newly diagnosed acute lymphoblastic leukemia (ALL). Dasatinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving dasatinib together with combination chemotherapy may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility and toxicity of an intensified chemotherapeutic regimen that incorporates dasatinib for treatment of children, adolescents, and young adults (up to age 30) with Philadelphia chromosome positive (Ph+) acute lymphoblastic leukemia (ALL).

II. To determine whether the intensification of tyrosine kinase inhibition through the addition of dasatinib in Induction (Days 15-28) and substitution of dasatinib for imatinib during post-Induction therapy, in the context of intensive cytotoxic therapy (according to AALL0031) and a good early response to therapy, will lead to a 3-year event-free survival (EFS) of at least 60% in patients with Ph+ ALL.

SECONDARY OBJECTIVES:

I. To determine whether the addition of dasatinib during Induction therapy (Days 15-28) will decrease levels of minimal residual disease (MRD) present at end of Induction therapy as compared with COG AALL0031.

II. To determine whether early intensified tyrosine kinase inhibitor (TKI) therapy will lower end-Consolidation MRD levels as compared to patients on COG AALL0031 that received imatinib in Consolidation Blocks 1 and 2 (Cohorts 3-5).

III. To determine the overall 3-year EFS rate for the whole cohort of Standard- and High-Risk patients treated with dasatinib.

IV. To determine the long-term effects of dasatinib on growth, development, and bone metabolism.

V. To assess BCR-ABL mutation status at time of diagnosis and progression/relapse.

OUTLINE: This is a multicenter study. Patients are stratified according to risk (standard risk vs high risk) at the end of consolidation therapy.

INDUCTION THERAPY (weeks 1-4): Patients receive initial induction therapy on days 1-14 prior to beginning the study. Patients then receive vincristine intravenously (IV) and daunorubicin hydrochloride* IV over 15 minutes on days 15 and 22; dasatinib orally (PO) once daily (QD) and prednisone PO (or methylprednisolone IV) twice daily (BID) on days 15-28; methotrexate intrathecally (IT) on day 29; and some patients receive methotrexate, hydrocortisone, and cytarabine IT on days 15 and 22. After completion of induction therapy, patients undergo bone marrow aspiration for evaluation of disease. Patients with M1 bone marrow and minimal residual disease (MRD) < 1% (standard-risk disease) proceed to block 1 consolidation therapy 1 week after completion of induction therapy or when blood counts recover (whichever occurs later). Patients with M2 or M3 bone marrow or MRD >= 1% (high-risk disease) proceed immediately to block 1 consolidation therapy, regardless of blood counts. Patients with clinically evident or biopsy-proven testicular leukemia at diagnosis that persists at the end of induction therapy undergo 12 fractions of testicular radiotherapy beginning within 4 days prior to starting block 1 consolidation therapy.

NOTE: *Patients who receive initial induction therapy on a DFCI Childhood ALL Consortium trial do not receive daunorubicin hydrochloride during induction therapy on this study.

CONSOLIDATION THERAPY:

BLOCK 1 CONSOLIDATION THERAPY: (weeks 6-8) Patients receive etoposide IV over 1 hour and ifosfamide IV over 1 hour on days 1-5, dasatinib PO on days 1-14 OR on days 1-21, and some patients receive methotrexate, hydrocortisone, and cytarabine IT on days 8 and 15. Patients also receive filgrastim (G-CSF) subcutaneously (SC) or IV QD beginning on day 6 and continuing until blood counts recover.

After completion of block 1 consolidation therapy, patients proceed to block 2 consolidation therapy.

BLOCK 2 CONSOLIDATION THERAPY: (weeks 9-11) Patients receive high-dose methotrexate IV continuously over 24 hours on day 1; leucovorin calcium PO or IV every 6 hours for 3 doses on days 2-3; methotrexate, hydrocortisone, and cytarabine IT on day 1; cytarabine IV over 3 hours every 12 hours for 4 doses on days 2 and 3; and dasatinib PO on days 1-14 OR on days 1-21. Patients also receive G-CSF SC or IV QD beginning on day 4 and continuing until blood counts recover. After completion of block 2 consolidation therapy and recovery of blood counts, patients undergo bone marrow aspiration for evaluation of disease. Patients with MRD < 0.01% (standard-risk disease) with a matched related donor and who are willing to undergo hematopoietic stem cell transplantation (HSCT) proceed to HSCT off study. Standard-risk patients without a suitable donor or those who elect not to undergo HSCT proceed to post-consolidation therapy. Patients with MRD >= 0.01% (high-risk disease) with a matched related or unrelated donor proceed to HSCT off study. High-risk patients without a suitable donor proceed to post-consolidation therapy.

POST-CONSOLIDATION THERAPY:

REINDUCTION BLOCK 1 THERAPY: (weeks 12-14) Patients receive vincristine IV on days 1, 8, and 15; daunorubicin hydrochloride IV over 15 minutes on days 1 and 2; cyclophosphamide IV over 1 hour every 12 hours for 4 doses on days 3 and 4; pegaspargase intramuscularly (IM) on day 4; methotrexate, hydrocortisone, and cytarabine IT on days 1 and 15; dexamethasone PO or IV BID on days 1-7 and 15-21; and dasatinib PO on days 1-14 OR on days 1-21. Patients also receive G-CSF SC or IV QD beginning on day 5 and continuing until blood counts recover.

After completion of reinduction block 1 therapy, patients proceed to intensification block 1 therapy.

INTENSIFICATION BLOCK 1 THERAPY: (weeks 15-23) Patients receive high-dose methotrexate IV continuously over 24 hours on day 1; leucovorin calcium PO or IV every 6 hours for 3 doses on days 2-3; methotrexate, hydrocortisone, and cytarabine IT on days 1 and 22; etoposide IV over 1 hour and cyclophosphamide IV over 1 hour on days 22-26; cytarabine IV over 3 hours every 12 hours for 4 doses on days 43 and 44; asparaginase IM on day 44; and dasatinib PO on days 1-14, 22-35, and 43-56 OR on days 1-63. Patients also receive G-CSF SC or IV QD beginning on day 27 and continuing until blood counts recover. After completion of intensification block 1 therapy, patients proceed to reinduction block 2 therapy.

REINDUCTION BLOCK 2 THERAPY: (weeks 24-26) Patients receive reinduction block 2 therapy as per reinduction block 1 therapy. After completion of reinduction block 2 therapy, patients proceed to intensification block 2 therapy.

INTENSIFICATION BLOCK 2 THERAPY: (weeks 27-35) Patients receive intensification block 2 therapy as per intensification block 1 therapy. After completion of intensification block 2 therapy, patients proceed to maintenance therapy.

MAINTENANCE THERAPY:

MAINTENANCE COURSES 1-4: (weeks 36-67) Patients receive high-dose methotrexate IV continuously over 24 hours on day 1; leucovorin calcium PO or IV every 6 hours for 3 doses on days 2-3; methotrexate, hydrocortisone, and cytarabine IT and vincristine IV on days 1 and 29; prednisone PO or IV BID on days 1-5 and 29-33; mercaptopurine PO on days 8-28; methotrexate PO on days 8, 15, and 22; etoposide IV over 1 hour and cyclophosphamide IV over 1 hour on days 29-33; and dasatinib PO on days 1-14 and 29-42 OR on days 1-56. Patients also receive G-CSF SC or IV QD beginning on day 34 and continuing until blood counts recover. Courses repeat every 56 days. After completion of maintenance courses 1-4, patients proceed to maintenance course 5.

MAINTENANCE COURSE 5: (weeks 68-75) Patients receive vincristine IV on days 1 and 29; prednisone PO or IV BID on maintenance courses 6-12.

MAINTENANCE COURSES 6-12: (weeks 76-131) Patients receive vincristine IV on days 1 and 29; prednisone PO or IV BID on days 1-5 and 29-33; mercaptopurine PO on days 1-56; methotrexate PO on days 1, 8, 15, 22, 29, 36, 43, and 50; and dasatinib PO on days 1-14 and 29-42 OR on days 1-56.

Courses repeat every 56 days. Patients long-term growth, development, and bone metabolism are assessed after completion of study therapy and then annually for 5 years.

After completion of study therapy, patients are followed up periodically for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed acute lymphoblastic leukemia (ALL)

  * Definitive evidence of BCR-ABL fusion (Philadelphia chromosome positive [PH+]) from an approved Children's Oncology Group (COG) cytogenetics laboratory
* Meets one of the following criteria:

  * Concurrent enrollment on Clusters of Orthologous Groups (COG)-AALL03B1 (or a successor trial) AND COG-AALL0232, COG-AALL0331, COG-AALL0434 or other front-line COG ALL clinical trial
  * Concurrent enrollment on COG-AALL03B1 (or a successor trial) AND scheduled to receive a 3 or 4-drug standard induction regimen
  * Concurrent enrollment on a Dana-Farber Cancer Institute (DFCI) Childhood ALL Consortium trial (or scheduled to be treated as per a DFCI Childhood ALL Consortium induction regimen)
* All patients must have definitive evidence of BCR-ABL fusion from an approved COG cytogenetics laboratory; patients may NOT have received Day 15 of Induction chemotherapy (or day 18 vincristine if enrolled on a DFCI Childhood ALL Consortium trial) prior to enrollment on AALL0622
* Patients must have a performance status of 0, 1 or 2 at completion of two weeks of Induction; use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70mL/min/1.73 m^2 or maximum serum creatinine based on age and gender as follows:

  * 0.4 mg/dL (for patients 1 to 5 months of age)
  * 0.5 mg/dL (for patients 6 to 11 months of age)
  * 0.6 mg/dL (for patients 1 year of age)
  * 0.8 mg/dL (for patients 2 to 5 years of age)
  * 1.0 mg/dL (for patients 6 to 9 years of age)
  * 1.2 mg/dL (for patients 10 to 12 years of age)
  * 1.5 mg/dL (males) or 1.4 mg/dL (females) (for patients 13 to 15 years of age)
  * 1.7 mg/dL (males) or 1.4 mg/dL (females) (for patients >= 16 years of age)
* Total bilirubin =< 1.5 times upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 2.5 times ULN for age
* Shortening fraction >= 27% by echocardiogram or ejection fraction >= 50% by gated radionuclide study
* No evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry > 94% at sea level if there is clinical indication for determination
* Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled; however, drugs that induce CYP3A4/5 (carbamazepine, oxcarbazepine, phenytoin, primidone, phenobarbital) should be avoided
* Patients will start AALL0622 therapy on day 15 of induction therapy (or day 18 if enrolled on a DFCI Childhood ALL Consortium trial); patients must have received the first 2 weeks of Induction therapy

Exclusion Criteria:

* Females of childbearing potential must have a negative pregnancy test; patients of childbearing potential must agree to use an effective birth control method
* Female patients who are lactating must agree to stop breast-feeding
* Patients with Down syndrome
* Patients with any clinically significant cardiovascular disease including the following:

  * Myocardial infarction or ventricular tachyarrhythmia within 6 months
  * Ejection fraction less than institutional normal
  * Major conduction abnormality (unless a cardiac pacemaker is present)

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2008-07-14 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William B Slayton, Principal Investigator — Children's Oncology Group
Locations (134):
- United States (118):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Harbor-University of California at Los Angeles Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (9):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- San Jorge Children's Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Tasian SK, Peters C. Targeted therapy or transplantation for paediatric ABL-class Ph-like acute lymphocytic leukaemia? Lancet Haematol. 2020 Dec;7(12):e858-e859. doi: 10.1016/S2352-3026(20)30369-0. No abstract available. PMID 33242441
- [Derived] Slayton WB, Schultz KR, Kairalla JA, Devidas M, Mi X, Pulsipher MA, Chang BH, Mullighan C, Iacobucci I, Silverman LB, Borowitz MJ, Carroll AJ, Heerema NA, Gastier-Foster JM, Wood BL, Mizrahy SL, Merchant T, Brown VI, Sieger L, Siegel MJ, Raetz EA, Winick NJ, Loh ML, Carroll WL, Hunger SP. Dasatinib Plus Intensive Chemotherapy in Children, Adolescents, and Young Adults With Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia: Results of Children's Oncology Group Trial AALL0622. J Clin Oncol. 2018 Aug 1;36(22):2306-2314. doi: 10.1200/JCO.2017.76.7228. Epub 2018 May 29. PMID 29812996

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Induction (Enzyme Inhibitor Therapy & Chemotherapy): See Detailed Description
  Asparaginase: Given IT
  Cyclophosphamide: Given IV
  Cytarabine: Given IT or IV
  Dasatinib: Given PO
  Daunorubicin Hydrochloride: Given IV
  Dexamethasone: Given IV or PO
  Etoposide: Given IV
  Filgrastim: Given IV or SC
  Hydrocortisone Sodium Succinate: Given IT
  Ifosfamide: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Leucovorin Calcium: Given IV or PO
  Mercaptopurine: Given PO
  Methotrexate: Given IT, PO, or IV
  Methylprednisolone: Given IV
  Pegaspargase: Given IM
  Prednisone: Given PO or IV
  Radiation Therapy: Some patients undergo cranial RT
  Vincristine Sulfate: Given IV
- Standard-risk: Based on Minimal Residual Disease, less than 1%.
- High-risk: Based on Minimal Residual Disease, great than or equal to 1%.
Period: Induction Period
Arm/Group | Treatment Induction (Enzyme Inhibitor Therapy & Chemotherapy) | Standard-risk | High-risk
Started | 63 | 0 | 0
Completed | 57 | 0 | 0
Not Completed | 6 | 0 | 0
Not completed — Did not meet eligibility criteria | 3 | 0 | 0
Not completed — Bone Marrow Transplant | 2 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Period: Risk Stratification Period
Arm/Group | Treatment Induction (Enzyme Inhibitor Therapy & Chemotherapy) | Standard-risk | High-risk
Started | 0 | 48 | 9
Completed | 0 | 33 | 1
Not Completed | 0 | 15 | 8
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Physician Decision | 0 | 2 | 1
Not completed — Bone marrow transplant | 0 | 9 | 7
Not completed — Disease progression or relapse | 0 | 2 | 0
Not completed — Development of second malignant neoplasm | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Since all patients were enrolled under induction therapy and later risk stratified, all patients are grouped under the treatment induction group, including the three ineligible patients.
Arm/Group | Treatment Induction (Enzyme Inhibitor Therapy & Chemotherapy)
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 56
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 9
  White | 45
  More than one race | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Event-Free Survival (EFS) of Patients With Standard-risk Disease Treated With Dasatinib in Combination With Intensified Chemotherapy
Description: Event-Free Survival (EFS) curves will be constructed using the Kaplan-Meier life table method with standard errors computed using the method of Peto and Peto. A 1-sided 95% confidence interval for EFS will be constructed.
Time Frame: At 3 years
Population: Patients with Philadelphia chromosome positive (Ph+) acute lymphoblastic leukemia (ALL).
Measure: Number (90% Confidence Interval); unit: Percent probability
Arm/Group | Treatment Induction (Enzyme Inhibitor Therapy & Chemotherapy) | Standard-risk | High-risk
Number analyzed (Participants) | 60 | 48 | 9
Percent probability | 79.8 [71.1 to 88.5] | 83.2 [74.1 to 92.2] | 66.7 [40.9 to 92.5]

2. Primary Outcome: Feasibility and Toxicity of an Intensified Chemotherapeutic Regimen Incorporating Dasatinib for Treatment of Children and Adolescents With Ph+ ALL Assessed by Examining Adverse Events
Description: Number of patients in safety cohort with dose limiting toxicity (DLT)(including treatment delay)
Time Frame: Weeks 3 through 23 of treatment (From week 3 Induction through Intensification Block 1)
Population: Patients with Philadelphia chromosome positive (Ph+) acute lymphoblastic leukemia (ALL)
Measure: Number; unit: Pts with DLTs
Groups:
- Treatment Induction (Enzyme Inhibitor Therapy & Chemotherapy): Feasibility measured by DLT rates in safety phase, Toxicities define DLTs and are summarized and reviewed to assess feasibility of administering the combination therapy with dasatinib
Arm/Group | Treatment Induction (Enzyme Inhibitor Therapy & Chemotherapy)
Number analyzed (Participants) | 12
Pts with DLTs | 1

3. Secondary Outcome: Contribution of Dasatinib on Minimal Residual Disease (MRD) After Induction Therapy
Description: Percent of patients MRD Positive (MRD > 0.01%) at End of Induction.
Time Frame: At the end of induction therapy (at 5 weeks)
Population: Patients with Philadelphia chromosome positive (Ph+) acute lymphoblastic leukemia (ALL).
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment Induction (Enzyme Inhibitor Therapy & Chemotherapy) | Standard-risk | High-risk
Number analyzed (Participants) | 59 | 48 | 9
Percentage of participants | 40.7 [30.8 to 51.4] | 29.2 [19.7 to 40.9] | 100.0 [73.1 to 100.0]
Statistical Analysis 1: Comparison: Treatment Induction (Enzyme Inhibitor Therapy & Chemotherapy); The a priori plan was to compare MRD positivity rate with that on a prior study, AALL0031 (n=72 Cohorts 1-5 of AALL0031 with 71% MRD positive). Out of 59 patients with end-Induction MRD on AALL0622, 40.7% were MRD positive. Per protocol, rates will be compared with a 2 sample Z-test of proportions, 1-sided test, alpha=5%; Test type: Superiority or Other; p < 0.001, Chi-squared; Chi-squared test equivalent to Z-test of proportions; Percentage = 40.7, 90% CI 2-sided [30.8 to 51.4]

4. Secondary Outcome: Percent of Patients MRD Positive (MRD > 0.01%) at End of Consolidation
Description: A 1-sample Z-test of proportions (alpha=5%, 1-sided test) will be used.
Time Frame: At end of consolidation (at 11 weeks)
Population: Patients with Philadelphia chromosome positive (Ph+) acute lymphoblastic leukemia (ALL).
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment Induction (Enzyme Inhibitor Therapy & Chemotherapy) | Standard-risk | High-risk
Number analyzed (Participants) | 57 | 48 | 9
Percentage of participants | 10.5 [5.3 to 19.3] | 0 [0.0 to 6.4] | 66.7 [39.6 to 96.1]
Statistical Analysis 1: Comparison: Treatment Induction (Enzyme Inhibitor Therapy & Chemotherapy); Test type: Superiority or Other; p = 0.13, Binomial Test; percentage = 10.5, 90% CI 2-sided [5.3 to 19.3] — The pre-specified threshold for the estimated percentage of MRD positivity at End Consolidation was set to 16%. Results show an upper bound on the (Agresti-Coull) confidence interval of 19.3%

5. Secondary Outcome: Overall EFS Rate for the Combined Cohort of Standard- and High-Risk Patients (Who Receive the Final Chosen Dose of Dasatinib)
Description: An event is defined as: Induction failure, relapse at any site, secondary malignancy, or death.
Time Frame: From the time entry on study to first event or date of last follow-up, assessed up to 7 years
Population: Included in the analysis are two patients who received the drug therapy but were not risk classified.
Measure: Number (90% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment Induction (Enzyme Inhibitor Therapy & Chemotherapy) | Standard-risk | High-risk
Number analyzed (Participants) | 60 | 48 | 9
percentage of patients | 79.8 [71.1 to 88.5] | 83.2 [74.1 to 92.2] | 66.7 [40.9 to 92.5]

ADVERSE EVENTS:
Description: SAE field contains NCI CTCAEs submitted via expedited reporting (NCI AdEERs / CAeRs). The AE field contains grade 3 and higher CTCAEs reported on study excluding those that were reported as SAEs.
Arm/Group | Treatment Induction (Enzyme Inhibitor Therapy & Chemotherapy) | Standard-risk | High-risk
Serious Adverse Events (participants affected / at risk) | 36/60 | 28/48 | 7/9
Other Adverse Events (participants affected / at risk) | 59/60 | 48/48 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Induction (Enzyme Inhibitor Therapy & Chemotherapy) (N=60) | Standard-risk (N=48) | High-risk (N=9)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 16 (23) | 11 (17) | 5 (6)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (5) | 2 (3) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 9 (11) | 6 (8) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 2 (2) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Confusion (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 2 (2) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 4 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 1 (1) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 (2) | 2 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 3 (3) | 1 (1)
Fever (General disorders) | 1 (1) | 1 (1) | 0 (0)
GGT increased (Investigations) | 2 (2) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (3) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (2)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (5) | 3 (3) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (4) | 2 (2) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 9 (12) | 6 (8) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 5 (6) | 4 (4) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 4 (5) | 4 (5) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
INR increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 7 (11) | 4 (6) | 2 (4)
Infusion related reaction (General disorders) | 1 (1) | 1 (1) | 0 (0)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (3) | 1 (2) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (3) | 1 (3) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (6) | 2 (4) | 1 (2)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Periorbital infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 2 (3) | 1 (1) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Personality change (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (5) | 2 (3) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (2) | 1 (2) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, spec (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 3 (3) | 3 (3) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 3 (6) | 2 (4) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Induction (Enzyme Inhibitor Therapy & Chemotherapy) (N=60) | Standard-risk (N=48) | High-risk (N=9)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 7 (7) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Acoustic nerve disorder NOS (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 31 (119) | 29 (114) | 2 (5)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 3 (3) | 2 (2) | 1 (1)
Anal mucositis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Anaphylaxis (Immune system disorders) | 5 (5) | 3 (3) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 23 (66) | 19 (61) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 5 (11) | 5 (11) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 20 (36) | 19 (35) | 1 (1)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 5 (7) | 3 (5) | 2 (2)
Bone infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (2) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 3 (8) | 2 (7) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (2) | 1 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 4 (5) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 9 (13) | 8 (12) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 6 (16) | 5 (15) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
External ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (4) | 2 (2) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 41 (148) | 36 (138) | 4 (9)
Fever (General disorders) | 4 (6) | 4 (6) | 0 (0)
Fibrinogen decreased (Investigations) | 4 (4) | 4 (4) | 0 (0)
GGT increased (Investigations) | 3 (5) | 3 (5) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (2) | 1 (2) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 5 (9) | 3 (7) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 13 (16) | 10 (13) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 5 (7) | 3 (3) | 2 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 (8) | 7 (7) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 9 (10) | 7 (8) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 29 (57) | 27 (51) | 1 (5)
Hyponatremia (Metabolism and nutrition disorders) | 14 (17) | 11 (14) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (7) | 2 (3) | 1 (4)
Hypotension (Vascular disorders) | 7 (8) | 7 (8) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 37 (99) | 34 (92) | 2 (6)
Infective myositis (Infections and infestations) | 1 (2) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 5 (7) | 5 (7) | 0 (0)
Lymphocyte count decreased (Investigations) | 8 (8) | 6 (6) | 2 (2)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 17 (24) | 16 (23) | 0 (0)
Musculoskeletal and connective tissue disorder - Ot (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 10 (23) | 9 (22) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 3 (3) | 3 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 41 (144) | 38 (140) | 2 (3)
Oral pain (Gastrointestinal disorders) | 1 (2) | 1 (2) | 0 (0)
Otitis media (Infections and infestations) | 5 (8) | 5 (8) | 0 (0)
Pain (General disorders) | 2 (3) | 2 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 2 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 8 (17) | 7 (16) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (17) | 9 (17) | 0 (0)
Personality change (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 33 (83) | 29 (79) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Psychosis (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (8) | 4 (7) | 1 (1)
Rectal mucositis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Ot (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (2) | 1 (2) | 0 (0)
Skin infection (Infections and infestations) | 9 (10) | 9 (10) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Small intestine infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (2) | 1 (2) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Trigeminal nerve disorder (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 3 (3) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (7) | 3 (7) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 10 (16) | 10 (16) | 0 (0)
White blood cell decreased (Investigations) | 24 (80) | 20 (75) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less